CLINICAL TRIAL: NCT00931645
Title: Randomized Phase III Trial Evaluating the Role of Autologous Stem Cell Transplantation in Previously Untreated Patients With Stage B and C Chronic Lymphocytic Leukemia
Brief Title: Autologous Stem Cell Transplantation in Chronic Lymphocytic Leukemia
Acronym: Auto-LLC 2001
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: Direction Générale de la Santé, France (Other)
Responsible Party: Laurent Sutton MD, SFGM-TC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFGMTC; PHRC
Record Dates: First submitted 2009-06-29; First posted 2009-07-02 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic lymphocytic leukemia,; autologous stem cell transplantation
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cisplatin; Dexamethasone; Cytarabine; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Complete responders (No Intervention): watch and wait policy
- arm 2: complete responders patients (Experimental): ABMT : TBI, 10 grays d-3-1 & cyclophosphamide 60 mg/sqm d-5-4
  Interventions: Procedure: Autologous stem cell transplantation
- Non CR patients arm 3 (Experimental): Rescue chemotherapy and ABMT (see arm 2)
  Interventions: Procedure: DHAP rescue and Autologous stem cell transplantation
- Non CR patients at random : arm 4 (Active Comparator): Rescue DHAP, F+C
  Interventions: Procedure: DHAP rescue and F+C

INTERVENTIONS:
Procedure: Autologous stem cell transplantation — TBI (10 grays, d-3-1), cyclophosphamide (60 mg/sqm d-5-4)
  Other Names: ABMT
  Arms: arm 2: complete responders patients
Procedure: DHAP rescue and Autologous stem cell transplantation — DHAP :IV cisplatin 100 mg/sqm d1, IV cytarabine 2 g/sqm d2,, IV dexamethasone 40 mg/sqm d1-4, TBI (10 grays d-3-1), cyclophosphamide (60 mg/sqm d-5-4)
  Other Names: cisplatin; dexamethasone; cytarabine
  Arms: Non CR patients arm 3
Procedure: DHAP rescue and F+C — DHAP :IV cisplatin 100 mg/sqm d1, IV Cytarabine 2 g/sqm d2, IV dexamethasone 40 mg/sqm d1-4, Followed by 3 monthly cycles with IV d1-3 fludarabine (25 mg/sqm) & cyclophosphamide (300 mg/sqm)
  Other Names: Fludarabine; Cyclophosphamide
  Arms: Non CR patients at random : arm 4

SUMMARY:
Phase III trial evaluating the role of autologous stem cell transplantation in previously untreated patients under 65 years with stage B and C B-cell chronic lymphocytic leukemia.

Endpoints of the trial :

* major : progression free survival at 3 years
* secondary : overall survival, tolerance, prognostic factors according to baseline clinical stage and biological characteristics (IgHv mutational status, expression of ZAP70 and CD38, cytogenetics).

DETAILED DESCRIPTION:
All registered patients will be treated with 6 monthly courses of chemotherapy. First three ones will be a CHOP regimen with half dosage of adriamycin, as previously published (Effectiveness of "CHOP" regimen in advanced untreated chronic lymphocytic leukemia. French Cooperative Group on Chronic Lymphocytic Leukemia. Lancet ; 1986, i : 1346-1349), followed by three subsequent courses with IV fludarabine (25 mg/sqm d1-5). Patients in CR (NCI, 1996, including CAT scan evaluation) will be then randomized to surveillance without additional treatment or autologous stem cell transplantation using peripheral stem cells collected after the three first courses of chemotherapy, and/or after the completion of the six courses when necessary. For patients not in CR after the six courses, a rescue regimen with the DHAP association ( cisplatin, 100 mg/sqm d1, cytarabine 2 g/sqm d2, dexamethasone 40 mg/sqm d1-4) will precede an additional stem cell collection if necessary, and patient will be randomized between autologous stem cell transplantation and three additional courses of an association of fludarabine (25 mg/sqm d1-3) and cyclophosphamide (300 mg/sqm d1-3). Conditioning regimen will associate TBI (10 grays, d -3-1) and cyclophosphamide (60 mg/sqm d-5-4).

Evaluation for response wil be performed before randomisation and two months after completion of therapy in each arm.

Follow-up data will be registered and monitored every three month during the first year, and then every six month. Criteria for evaluation of response will use the NCI system (1996).

ELIGIBILITY:
Inclusion Criteria:

* patients with stage B & C CLL, 18- 65 years.
* previously untreated
* given written informed consent

Exclusion Criteria:

* Childbearing women
* OMS Performance status > 2
* Binet stage A
* Autoimmune hemolytic anemia
* Active or previous (< 5 years) malignant disease, except cutaneous cell carcinoma.
* Previous CLL treatment
* HIV seropositivity
* Abnormal renal or liver function tests (creatinine > 1,5N, transaminases > 2N, bilirubin > 1,5N)
* Cardiac failure (ejection fraction < 50%)
* Lung disease or perturbed ventilation tests

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2001-04; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 3 year

SECONDARY OUTCOMES:
Overall survival, response after completion of scheduled treatment, tolerance and adverse events, quality of life, prognostic factors for response and survival. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Sutton Laurent, MD, Principal Investigator — Hospital Victor Dupouy Argenteuil, France; Leporrier Michel, MD, Study Chair — CaenUH, France
Locations (1):
- DBIM Hopital Saint Louis, Paris, France